CLINICAL TRIAL: NCT05969340
Title: Detecting Otoconia Using Ultra-high Resolution CT-imaging in Patients With Posterior Canal Benign Paroxysmal Positional Vertigo
Brief Title: Detecting Otoconia With CT-Scan
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is still in the planning stage, undergoing protocol reconsideration.
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Responsible Party: Principal Investigator, Ali Melliti, Audiologist, PhD Candidate, Academisch Ziekenhuis Maastricht
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NL 83124.068.22
Record Dates: First submitted 2023-07-14; First posted 2023-08-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: BPPV
Keywords: BPPV; Otoconia; ultra-high resolution CT-imaging

STUDY DESIGN:
Intervention Model Description: There are 2 groups involved:
  * The experimental group
  * The control group
Who Masked: Outcomes Assessor
Masking Description: The radiologist assessing the CT imaging will be blinded to which participants have positive posterior canal BPPV.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patient diagnosed with Posterior canal BPPV
  Interventions: Diagnostic Test: ultra-high-resolution CT-scan
- Control group (Placebo Comparator): Patient who are scheduled for CT-imaging as part of standard clinical routine and do not have BPPV
  Interventions: Diagnostic Test: ultra-high-resolution CT-scan

INTERVENTIONS:
Diagnostic Test: ultra-high-resolution CT-scan — Use of ultra-high-resolution CT-scan to detect otoconia in the posterior canal BPPV

SUMMARY:
Benign Paroxysmal Positional Vertigo (BPPV) is a benign inner ear disease that causes the patient to experience short episodes of vertigo when there are changes in head position. The current theory on the causes of BPPV is the displacement of the otoconia from the otolith organ to the semicircular canal organs. BPPV's current treatments consist of repositioning maneuvers to readjust the location of the otoconia back to its original place. Even though the treatments are highly successful in many cases, this study, if proven successful, will help confirm this theory and will help diagnose complicated cases where BPPV is recurrent and treatment has been unsuccessful.

DETAILED DESCRIPTION:
Benign Paroxysmal Positional Vertigo (BPPV) is a benign inner ear disease that causes the patient to experience vertigo when there are changes in head position. The prevalence is estimated to account for 20-30% of all vertigo diagnoses in a specialized clinic (von Brevern et al., 2007). The current theory on the cause of BPPV is the displacement of otoconia from the otolith organ to the semicircular canal organs due to gravitational forces.

Current treatments for BPPV consist of repositioning maneuvers to readjust the location of the otoconia back to its original place (von Brevern et al., 2015). Even though the treatment is highly successful in many cases patients still have recurrent (26%) or persistent (4%) symptoms (Dorigueto et al., 2009), and objective confirmation of the disease is warranted. Until now, visualization and confirmation of the presence of otoliths have not been successful in clinical practice. This is largely due to the very small size of the otoliths in a small inner ear structure, requiring sensitive and ultra-high-resolution imaging.

In 2021, a study was performed in Japan using 3 Dimensional Computed Tomography (3D CT) scans to detect the otoconia inside the horizontal canal. It compared scans of people with BPPV in the horizontal canal and healthy individuals (Yamane et al., 2021). The authors were able to visualize otoconia-like substance inside the canal in all 10 out of 10 affected patients and 6 out of 10 of the healthy participants in at least one ear (Yamane et al., 2021). In this study, the investigators will image the patients temporal bone with an ultra-high-resolution CT-scan (Benson et al.2022). They will focus on imaging the posterior canal for BPPV, and compare it with the imaging of individuals who do not have BPPV. In addition, they will compare the imaging of the canal pre and post-treatment using the Epley maneuver.

ELIGIBILITY:
Inclusion Criteria:

Experimental Group:

* Diagnosed with Posterior canal BPPV.
* Age 18 or older.
* Clear nystagmus consistent with canal direction and stimulation.
* Mild or greater complaints (none, mild, moderate, severe).
* Crescendo decrescendo nystagmus pattern.
* Slow phase eye velocity ≥ 15 deg/sec.

Control Group:

* Scheduled for CI implantation CT scan.
* Age 18 or older.

Exclusion Criteria:

Experimental Group:

* Anterior or lateral canal BPPV.
* Inability to undergo CRM and DH maneuvers.
* Central vestibular disorders.
* Multi-canal BPPV or subjective BPPV.
* Pregnancy.

Control Group:

* BPPV, central vestibular disorders, multicanal BPPV, subjective BPPV.
* Ossifying labyrinthitis, DFNA9, obstructive vestibular schwannoma on MRI.
* Normal VHIT or history of meningitis.
* Pregnancy or other vestibular pathologies.
* Past history of BPPV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Visualisation of presence or absence of otoconia in the posterior semicircular canal by comparing patient with confirmed BPPV symptoms compared to control subjects without BPPV | up to 1 hour
  The presence or absence of otoconia in the posterior semicircular canal will be assessed qualitatively and semi-quantitatively using the CT parameters for BPPV patients, and the radiological images will be compared to those of control subjects.

SECONDARY OUTCOMES:
Visualization of the presence or absence of otoconia in patients with confirmed Benign Paroxysmal Positional Vertigo (BPPV) symptoms before and after a repositioning procedure. | up to 1 hour
  Change in position of the otoconia will be assessed qualitatively and semi-quantitively using the CT parameters in BPPV patients by comparing the radiological images before and after repositioning maneuver (Epley)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] von Brevern M, Radtke A, Lezius F, Feldmann M, Ziese T, Lempert T, Neuhauser H. Epidemiology of benign paroxysmal positional vertigo: a population based study. J Neurol Neurosurg Psychiatry. 2007 Jul;78(7):710-5. doi: 10.1136/jnnp.2006.100420. Epub 2006 Nov 29. PMID 17135456
- [Background] von Brevern M, Bertholon P, Brandt T, Fife T, Imai T, Nuti D, Newman-Toker D. Benign paroxysmal positional vertigo: Diagnostic criteria. J Vestib Res. 2015;25(3-4):105-17. doi: 10.3233/VES-150553. PMID 26756126
- [Background] Dorigueto RS, Mazzetti KR, Gabilan YP, Gananca FF. Benign paroxysmal positional vertigo recurrence and persistence. Braz J Otorhinolaryngol. 2009 Jul-Aug;75(4):565-72. doi: 10.1016/s1808-8694(15)30497-3. PMID 19784427
- [Background] Yamane H, Konishi K, Anniko M. Visualization of horizontal canal benign paroxysmal positional vertigo using 3DCT imaging and its assessment. Acta Otolaryngol. 2021 May;141(5):482-489. doi: 10.1080/00016489.2021.1892822. Epub 2021 Mar 29. PMID 33781168
- [Background] Rajendran K, Voss BA, Zhou W, Tao S, DeLone DR, Lane JI, Weaver JM, Carlson ML, Fletcher JG, McCollough CH, Leng S. Dose Reduction for Sinus and Temporal Bone Imaging Using Photon-Counting Detector CT With an Additional Tin Filter. Invest Radiol. 2020 Feb;55(2):91-100. doi: 10.1097/RLI.0000000000000614. PMID 31770297
- [Background] Benson JC, Rajendran K, Lane JI, Diehn FE, Weber NM, Thorne JE, Larson NB, Fletcher JG, McCollough CH, Leng S. A New Frontier in Temporal Bone Imaging: Photon-Counting Detector CT Demonstrates Superior Visualization of Critical Anatomic Structures at Reduced Radiation Dose. AJNR Am J Neuroradiol. 2022 Apr;43(4):579-584. doi: 10.3174/ajnr.A7452. Epub 2022 Mar 24. PMID 35332019